CLINICAL TRIAL: NCT00265083
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, a Fully Human Anti-TNFalpha MonoclonalAntibody, Administered Subcutaneously, in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study of the Safety and Efficacy of Golimumab in Subjects With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006337; C0524T09 (Other: Centocor)
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2009-07-13 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Spondylitis, Ankylosing
Keywords: Spondylitis; subcutaneous injection; Bechterew's Disease; Spondyloarthritis; Spondyloarthropathy
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylitis; Spondylarthritis; Spondylarthropathies | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 003 (Experimental): golimumab 100 mg sc injections every 4 wks from wk 0 up to 5 yrs
  Interventions: Biological: golimumab
- 001 (Placebo Comparator): Golimumab (CNTO 148); placebo SC injections every 4 wks thru wk 20 (unless early escape at wk 16);golimumab - if early escape, 50mg sc inj every 4wks from wk 16 up to 5yrs ;golimumab -50mg sc injection beginning wk 24 up to 5 yrs (unless early escape); golimumab- Dr's discretion after unblinding, dose adjust from 50 to 100mg
  Interventions: Biological: Golimumab (CNTO 148); placebo
- 002 (Experimental): golimumab 50 mg sc injs every 4wks from wk 0 thru 5yrs (unless early escape at wk 16); golimumab - If early escape, 100mg sc injections every 4 wks beginning wk 16 up to 5 yrs ; golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100mg
  Interventions: Biological: golimumab

INTERVENTIONS:
Biological: golimumab — 100 mg sc injections every 4 wks from wk 0 up to 5 yrs
  Arms: 003
Biological: Golimumab (CNTO 148); placebo — SC injections every 4 wks thru wk 20 (unless early escape at wk 16);golimumab - if early escape, 50mg sc inj every 4wks from wk 16 up to 5yrs ;golimumab -50mg sc injection beginning wk 24 up to 5 yrs (unless early escape); golimumab- Dr's discretion after unblinding, dose adjust from 50 to 100mg
  Arms: 001
Biological: golimumab — 50 mg sc injs every 4wks from wk 0 thru 5yrs (unless early escape at wk 16); golimumab - If early escape, 100mg sc injections every 4 wks beginning wk 16 up to 5 yrs ; golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100mg
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of subcutaneous injections (under the skin) of golimumab for the treatment of active ankylosing spondylitis [AS(arthritis of the spine)]. Efficacy will be measured by reduction in the signs and symptoms of active AS, including effects on back pain and stiffness, physical function, range of motion in the spine, quality of life, and rate of spine damage or fusion on x-ray.

DETAILED DESCRIPTION:
Anti-tumor necrosis factor (TNF) agents have been shown to be effective treatment for patients with active ankylosing spondylitis (arthritis of the spine) who have not responded to conventional therapy. Golimumab is a new anti-TNFa agent. This is a multicenter, randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled, parallel group study comparing safety and efficacy of golimumab 50mg, golimumab 100mg, and placebo subcutaneous (under the skin) injections administered every 4 weeks, in patients with active AS. The total duration of treatment is approximately 5 years. In the first portion of the study, some patients will be randomly assigned to receive placebo treatment through the Week 20 injection; others will be assigned to golimumab 50mg or golimumab 100mg groups through the Week 20 injection. There is an "early escape" at Week 16 in the study whereby patients who meet criteria for having little improvement in their AS symptoms will be switched to golimumab if they were on placebo, or have the golimumab dose increased if they were originally assigned to the golimumab 50mg group. At Week 24, the placebo group patients will switch to golimumab 50mg injections, and all patients will continue receiving in a blinded manner either 50 or 100mg golimumab injections every 4 weeks until the first 104 weeks of data are fully collected on all the patients (database lock). After this 104-week database lock, everyone will be unblinded to the golimumab dose, and continue to receive golimumab treatment through Week 252 as part of a long-term extension phase of the study, with options for adjusting concomitant AS medications and/or increasing the dose of golimumab. The study hypothesis is that golimumab will be more effective than placebo in treating the signs and symptoms of AS, as measured by the ASsessment in Ankylosing Spondlitis (ASAS) 20 response criteria . Golimumab 50mg, Golimumab 100mg, or placebo injected under the skin every 4 weeks at Weeks 0, 4, 8, 12, 16, and 20, followed by injections of either Golimumab 50mg or Golimumab 100mg every 4 weeks for approximately 5 years total duration from the time of the first study agent injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "Definite AS" (arthritis of the spine) as defined by the modified New York criteria, for at least 3 months prior to first dose of study drug
* Symptoms of active disease at screening and at baseline visits, as evidenced by both a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of >= 4, and a Total Back Pain score of >= 4 (each on a scale of 0 to 10cm)
* Inadequate response to 3 months of continuous therapy with maximal recommended doses of NSAIDs, or else unable to receive a full 3 months of maximal NSAID therapy because of intolerance, toxicity, or contraindications to non-steroidal anti-inflammatory drugs (NSAIDs)
* Stable doses of methotrexate, sulfasalazine, hydroxychloroquine, low-dose corticosteroids, and NSAIDs are permitted.

Exclusion Criteria:

* Patients cannot have complete ankylosis of the spine
* No prior treatment with biologic anti-TNF agents (infliximab, etanercept, adalimumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (39):
- United States (11):
  - Paradise Valley, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Ormond Beach, Florida
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Houston, Texas
  - Edmonds, Washington
  - Seattle, Washington
  - Brookfield, Wisconsin
  - La Crosse, Wisconsin
- Belgium (3):
  - Brussels
  - Diepenbeek
  - Leuven
- Canada (7):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Toronto, Ontario
  - Sainte-Foy, Quebec
- Finland (2):
  - Helsinki
  - Rauma
- Nantes Cedex 01 N/A, France
- Germany (7):
  - Bad Nauheim
  - Baden-Baden
  - Berlin
  - Erlangen
  - Hanover
  - Herne
  - München
- Netherlands (2):
  - Maastricht
  - Nijmegen
- South Korea (3):
  - Busan
  - Pusan
  - Seoul
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taoyuan District

REFERENCES:
- [Derived] Leu JH, Adedokun OJ, Gargano C, Hsia EC, Xu Z, Shankar G. Immunogenicity of golimumab and its clinical relevance in patients with rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. Rheumatology (Oxford). 2019 Mar 1;58(3):441-446. doi: 10.1093/rheumatology/key309. PMID 30412238
- [Derived] Inman RD, Baraliakos X, Hermann KA, Braun J, Deodhar A, van der Heijde D, Xu S, Hsu B. Serum biomarkers and changes in clinical/MRI evidence of golimumab-treated patients with ankylosing spondylitis: results of the randomized, placebo-controlled GO-RAISE study. Arthritis Res Ther. 2016 Dec 28;18(1):304. doi: 10.1186/s13075-016-1200-1. PMID 28031053
- [Derived] Kay J, Fleischmann R, Keystone E, Hsia EC, Hsu B, Zhou Y, Goldstein N, Braun J. Five-year Safety Data from 5 Clinical Trials of Subcutaneous Golimumab in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, and Ankylosing Spondylitis. J Rheumatol. 2016 Dec;43(12):2120-2130. doi: 10.3899/jrheum.160420. Epub 2016 Nov 1. PMID 27803138
- [Derived] Braun J, Baraliakos X, Hermann KG, Xu S, Hsu B. Serum C-reactive Protein Levels Demonstrate Predictive Value for Radiographic and Magnetic Resonance Imaging Outcomes in Patients with Active Ankylosing Spondylitis Treated with Golimumab. J Rheumatol. 2016 Sep;43(9):1704-12. doi: 10.3899/jrheum.160003. Epub 2016 Jul 15. PMID 27422890
- [Derived] Braun J, Baraliakos X, Hermann KG, Xu S, Hsu B. Serum Vascular Endothelial Growth Factor Levels Lack Predictive Value in Patients with Active Ankylosing Spondylitis Treated with Golimumab. J Rheumatol. 2016 May;43(5):901-6. doi: 10.3899/jrheum.150897. Epub 2016 Mar 1. PMID 26932345
- [Derived] Deodhar A, Braun J, Inman RD, van der Heijde D, Zhou Y, Xu S, Han C, Hsu B. Golimumab administered subcutaneously every 4 weeks in ankylosing spondylitis: 5-year results of the GO-RAISE study. Ann Rheum Dis. 2015 Apr;74(4):757-61. doi: 10.1136/annrheumdis-2014-205862. Epub 2014 Nov 11. PMID 25387477
- [Derived] van der Heijde D, Braun J, Deodhar A, Inman RD, Xu S, Mack ME, Hsu B. Comparison of three enthesitis indices in a multicentre, randomized, placebo-controlled trial of golimumab in ankylosing spondylitis (GO-RAISE). Rheumatology (Oxford). 2013 Feb;52(2):321-5. doi: 10.1093/rheumatology/kes251. Epub 2012 Sep 28. PMID 23024015
- [Derived] van der Heijde D, Deodhar A, Inman RD, Braun J, Hsu B, Mack M. Comparison of three methods for calculating the Bath Ankylosing Spondylitis Metrology Index in a randomized placebo-controlled study. Arthritis Care Res (Hoboken). 2012 Dec;64(12):1919-22. doi: 10.1002/acr.21771. PMID 22740380
- [Derived] Deodhar A, Braun J, Inman RD, Mack M, Parasuraman S, Buchanan J, Hsu B, Gathany T, van der Heijde D. Golimumab reduces sleep disturbance in patients with active ankylosing spondylitis: results from a randomized, placebo-controlled trial. Arthritis Care Res (Hoboken). 2010 Sep;62(9):1266-71. doi: 10.1002/acr.20233. PMID 20506403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 356 patients were randomly assigned to treatment groups at 42 sites (17 in North America, 16 in Europe and 9 in Asia). Consent was obtained from the first patient on 13 Dec 2005. The last patient completed the final visit of the 24-week reporting period on 15 May 2007. The last patient completed the final visit of the 5-year period on 17 Jan 2012.
Groups:
- Group 1: Placebo: Placebo SC injections every 4 weeks (wks) from Week (Wk) 0 thru Wk 20 (unless early escape at Wk 16); golimumab - if early escape, 50 mg SC every 4 wks from Wk 16 up to 5 yrs; golimumab - 50 mg SC beginning Wk 24 up to 5 yrs (unless early escape); golimumab- Dr's discretion after unblinding, dose adjust from 50 to 100 mg.
- Group 2: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 wks from Wk 0 thru 5 yrs (unless early escape at Wk 16); golimumab - If early escape, 100 mg SC every 4 wks beginning Wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100 mg.
- Group 3: Golimumab 100 mg: Golimumab 100 mg SC injections every 4 wks from Wk 0 up to 5 yrs.
Period: Overall Study
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg
Started | 78 | 138 (One patient did not receive study agent.) | 140
Completed | 61 | 96 (One patient did not receive study agent.) | 98
Not Completed | 17 | 42 | 42
Not completed — Adverse Event | 5 | 13 | 15
Not completed — Lost to Follow-up | 3 | 4 | 4
Not completed — Unsatisfactory therapeutic effect | 8 | 13 | 14
Not completed — Other | 1 | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Group I: Placebo: Placebo SC injections every 4 weeks (wks) from Week (Wk) 0 thru Wk 20 (unless early escape at Wk 16); golimumab - if early escape, 50 mg SC every 4 wks from Wk 16 up to 5 yrs; golimumab - 50 mg SC beginning Wk 24 up to 5 yrs (unless early escape); golimumab- Dr's discretion after unblinding, dose adjust from 50 to 100 mg.
- Group II: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 wks from Wk 0 thru 5 yrs (unless early escape at Wk 16); golimumab - If early escape, 100 mg SC every 4 wks beginning Wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100 mg.
- Group III: Golimumab 100 mg: Golimumab 100 mg SC injections every 4 wks from Wk 0 up to 5 yrs.
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Total
Number analyzed (Participants) | 78 | 138 | 140 | 356
Age Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.71) | 39.2 (12.46) | 38.6 (11.30) | 39.3 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 36 | 42 | 101
  Male | 55 | 102 | 98 | 255

OUTCOME MEASURES:

1. Primary Outcome: Assessment in Ankylosing Spondylitis 20 Responders at Week 14
Description: Number of patients who achieved a 20% improvement and at least 1 absolute improvement on a 0 to 10 cm scale from baseline to Week 14 in at least 3 of the 4 domains: patient global, total back pain, function or inflammation.
Time Frame: Week 14
Population: Intent to treat (ITT). Patients considered non-responder if used any pre-specified prohibited medications or discontinued subcutaneous (SC) study agent due to lack of efficacy. Missing ASAS components at Week 14 were imputed by Last Observation Carried Forward (LOCF) unless all ASAS components are missing in which case considered non-responders.
Measure: Number; unit: Participants
Groups:
- Combined: Groups II & III: Combines Group II (golimumab 50 mg) and Group III (golimumab 100 mg).
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Groups II & III
Number analyzed (Participants) | 78 | 138 | 140 | 278
Participants | 17 | 82 | 84 | 166
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Groups II & III; Null hypothesis: No difference in ASAS 20 response comparing Groups I vs II and Groups I vs III. The sample size of 75 patients (pts) in placebo and 135 pts per active group will provide >=99% power to detect a difference in ASAS 20 response between treatment groups at alpha=0.05, assuming 50% of pts with screening CRP<1.5mg/dL, and the difference in ASAS 20 response of 10-27.5% in pts with screening CRP<1.5mg/dL and 32.5-45% in pts with screening CRP>=1.5mg/dL, between Groups I vs II or III; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The positive test is defined if the comparison between combined golimumab and placebo is significant (p-value <0.05), and at least one of the pair-wise comparisons is also significant (p-value <0.05); Cochran-Mantel-Haenszel with stratification: screening CRP level (<=1.5mg/dL, >1.5mg/dL)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with stratification: screening CRP level (<=1.5mg/dL, >1.5mg/dL)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with stratification: screening CRP level (<=1.5mg/dL, >1.5mg/dL)

2. Secondary Outcome: Assessment in Ankylosing Spondylitis 20 Responders at Week 24
Description: Number of patients who achieved a 20% improvement and at least 1 absolute improvement on a 0 to 10 cm scale from baseline to Week 24 at least 3 of the 4 domains: patient global, total back pain, function or inflammation.
Time Frame: Week 24
Population: ITT. Patients (pts) considered non-responder if used any pre-specified prohibited medications or discontinued SC study agent due to lack of efficacy. Missing ASAS components were imputed by LOCF unless all ASAS components are missing in which case considered non-responders. Wk 16 ASAS response was used for pts with change in study treatment.
Measure: Number; unit: P a r t i c ip an t s
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Groups II & III
Number analyzed (Participants) | 78 | 138 | 140 | 278
P a r t i c ip an t s | 18 | 77 | 92 | 169
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Groups II & III; Null hypothesis: No difference in ASAS 20 response comparing Groups I vs. II and Groups I vs. III; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel with stratification: screening CRP level (<=1.5mg/dL, >1.5mg/dL)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Null hypothesis: no difference in ASAS 20 response between Group II and Group I; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with stratification: screening CRP level (<=1.5mg/dL, >1.5mg/dL)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Null hypothesis: no difference in ASAS 20 response between Group III and Group I; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with stratification: screening CRP level (<=1.5mg/dL, >1.5mg/dL)

3. Secondary Outcome: Summary of Change From Baseline in Bath Ankylosing Spondylitis Functional Index at Week 14
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) is calculated as the mean of 10 VAS, each of length 0 to 10 cm. Eight of the scales relate to functional capacity of patients while the other 2 relate to a patient's ability to cope with everyday life. Change from baseline is Wk 14 value minus baseline value.
Time Frame: From Baseline to Week 14
Population: Intent to treat (ITT). Patients considered non-change from baseline in BASFI if used any pre-specified prohibited medications or discontinued SC study agent due to lack of efficacy. Missing value of change from baseline in BASFI at Week 14 was imputed by Last Observation Carried Forward (LOCF).
Measure: Median (Inter-Quartile Range); unit: Change from baseline in BASFI Index
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Groups II & III
Number analyzed (Participants) | 78 | 138 | 140 | 278
Change from baseline in BASFI Index | 0.095 [-1.050 to 1.120] | -1.375 [-3.130 to -0.120] | -1.495 [-2.985 to -0.060] | -1.420 [-3.070 to -0.080]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Groups II & III; Null hypothesis: No difference in change from baseline in BASFI comparing Groups I vs. II and Groups I vs. III; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores — [p-value comment as in outcome 1, analysis 1]; ANOVA on van der Waerden normal scores with 2 factors: treatment group and screening C-reactive protein (CRP) level
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Null hypothesis: no difference in BASFI between Group II and Group I; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; ANOVA on van der Waerden normal scores with 2 factors: treatment group and screening C-reactive protein (CRP) level
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Null hypothesis: no difference in BASFI between Group III and Group I; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; ANOVA on van der Waerden normal scores with 2 factors: treatment group and screening C-reactive protein (CRP) level

4. Secondary Outcome: Summary of Change From Baseline in Bath Ankylosing Spondylitis Metrology Index at Week 14
Description: The Bath Ankylosing Spondylitis Metrology Index (BASMI) is the sum of scores comprised of 5 measures (0=mild, 1=moderate & 2=severe): Tragus-to-wall; Lumbar flexion; Cervical rotation; Lumbar side flexion; Intermalleolar distance. BASMI ranges from 0 to 10. Change from baseline is Wk 14 value minus baseline value.
Time Frame: From Baseline to Week 14
Population: Intent to treat (ITT). Patients considered non-change from baseline in BASMI if used any pre-specified prohibited medications or discontinued SC study agent due to lack of efficacy. Missing value of change from baseline in BASMI at Week 14 was imputed by Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Change from baseline in BASMI Index
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Groups II & III
Number analyzed (Participants) | 78 | 138 | 140 | 278
Change from baseline in BASMI Index | -0.28 (1.015) | -0.36 (1.112) | -0.49 (1.296) | -0.43 (1.208)
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Groups II & III; Null hypothesis: No difference in change from baseline in BASMI comparing Groups I vs. II and Groups I vs. III; Test type: Superiority or Other; p = 0.288, ANOVA on van der Waerden normal scores — The positive test is defined if the comparison between combined golimumab and placebo is significant at the 0.05, and at least one of the pair-wise comparisons is also significant at the 0.05; ANOVA on van der Waerden normal scores with 2 factors: treatment group and screening C-reactive protein (CRP) level
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Null hypothesis: no difference in BASMI between Group II and Group I; Test type: Superiority or Other; p = 0.444, ANOVA on van der Waerden normal scores; ANOVA on van der Waerden normal scores with 2 factors: treatment group and screening C-reactive protein (CRP) level
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Null hypothesis: no difference in BASMI between Group III and Group I; Test type: Superiority or Other; p = 0.247, ANOVA on van der Waerden normal scores; ANOVA on van der Waerden normal scores with 2 factors: treatment group and screening C-reactive protein (CRP) level

ADVERSE EVENTS:
Time Frame: Up to 5 years (end of study)
Description: The number of participants reported at risk for adverse events (AEs) in each treatment (tx) group is based on actual tx received during the study and may differ from the number of participants who started tx in the study. Participants may be counted more than once in the analysis of AEs if they received tx at more than one dose level in the study.
Groups:
- Group 1: Golimumab 50 mg: Subjects who were treated with Golimumab and received Golimumab 50 mg injections only.
- Group 2: Golimumab 100 mg: Subjects who were treated with Golimumab and received Golimumab 100 mg injections only.
- Group 3: Golimumab 50 and 100 mg: Subjects who were treated with Golimumab and received at least one injection of both Golimumab 50 mg and Golimumab 100 mg.
Arm/Group | Group 1: Golimumab 50 mg | Group 2: Golimumab 100 mg | Group 3: Golimumab 50 and 100 mg
Serious Adverse Events (participants affected / at risk) | 27/158 | 26/118 | 19/77
Other Adverse Events (participants affected / at risk) | 147/158 | 113/118 | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg (N=158) | Group 2: Golimumab 100 mg (N=118) | Group 3: Golimumab 50 and 100 mg (N=77)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1
Hypertensive Heart Disease (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Malocclusion (Gastrointestinal disorders) | 1 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 2 | 0
Device Occlusion (General disorders) | 0 | 1 | 0
Generalised Oedema (General disorders) | 0 | 0 | 1
Biliary Colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 1
Bursitis Infective (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cellulitis Staphylococcal (Infections and infestations) | 0 | 0 | 1
Clostridial Infection (Infections and infestations) | 1 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 1 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 1 | 0
Lyme Disease (Infections and infestations) | 0 | 1 | 0
Otitis Media Chronic (Infections and infestations) | 0 | 1 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Post Procedural Infection (Infections and infestations) | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Face Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Prognathism (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1
Multiple Sclerosis (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Alcohol Abuse (Psychiatric disorders) | 0 | 1 | 0
Bipolar I Disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 2
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pregnancy of Partner (Social circumstances) | 0 | 1 | 0
Female Sterilisation (Surgical and medical procedures) | 1 | 0 | 0
Aortic Dissection (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg (N=158) | Group 2: Golimumab 100 mg (N=118) | Group 3: Golimumab 50 and 100 mg (N=77)
Dry Eye (Eye disorders) | 1 | 3 | 4
Iritis (Eye disorders) | 7 | 7 | 3
Uveitis (Eye disorders) | 7 | 10 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 5 | 5
Abdominal Pain (Gastrointestinal disorders) | 8 | 4 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 0 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 12 | 9 | 5
Dental Caries (Gastrointestinal disorders) | 2 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 16 | 11
Dyspepsia (Gastrointestinal disorders) | 10 | 11 | 2
Gastritis (Gastrointestinal disorders) | 8 | 4 | 1
Nausea (Gastrointestinal disorders) | 16 | 24 | 9
Toothache (Gastrointestinal disorders) | 3 | 7 | 3
Vomiting (Gastrointestinal disorders) | 9 | 8 | 4
Chest Pain (General disorders) | 7 | 4 | 5
Fatigue (General disorders) | 25 | 30 | 10
Injection Site Erythema (General disorders) | 8 | 12 | 10
Injection Site Swelling (General disorders) | 3 | 3 | 5
Oedema Peripheral (General disorders) | 8 | 7 | 4
Pyrexia (General disorders) | 13 | 11 | 4
Hepatic Steatosis (Hepatobiliary disorders) | 3 | 8 | 2
Seasonal Allergy (Immune system disorders) | 4 | 4 | 4
Bronchitis (Infections and infestations) | 17 | 12 | 10
Cellulitis (Infections and infestations) | 7 | 6 | 2
Ear Infection (Infections and infestations) | 2 | 7 | 1
Gastroenteritis (Infections and infestations) | 9 | 8 | 2
Gastroenteritis Viral (Infections and infestations) | 1 | 6 | 2
Herpes Zoster (Infections and infestations) | 3 | 4 | 6
Influenza (Infections and infestations) | 10 | 13 | 10
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 4 | 4
Nasopharyngitis (Infections and infestations) | 49 | 44 | 27
Oral Herpes (Infections and infestations) | 8 | 5 | 6
Pharyngitis (Infections and infestations) | 9 | 7 | 3
Rhinitis (Infections and infestations) | 9 | 6 | 4
Sinusitis (Infections and infestations) | 18 | 19 | 13
Tooth Abscess (Infections and infestations) | 4 | 4 | 4
Tooth Infection (Infections and infestations) | 6 | 7 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 60 | 42 | 26
Urinary Tract Infection (Infections and infestations) | 6 | 13 | 7
Vaginal Infection (Infections and infestations) | 2 | 0 | 4
Viral Infection (Infections and infestations) | 1 | 1 | 4
Vulvovaginal Mycotic Infection (Infections and infestations) | 3 | 7 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 4 | 6
Laceration (Injury, poisoning and procedural complications) | 2 | 8 | 3
Ligament Sprain (Injury, poisoning and procedural complications) | 9 | 4 | 1
Alanine Aminotransferase Increased (Investigations) | 21 | 20 | 5
Aspartate Aminotransferase Increased (Investigations) | 14 | 12 | 6
Blood Glucose Increased (Investigations) | 2 | 5 | 4
Weight Increased (Investigations) | 7 | 7 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 6 | 1
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 9 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 28 | 23
Back Pain (Musculoskeletal and connective tissue disorders) | 36 | 31 | 16
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 5 | 5 | 6
Joint Swelling (Musculoskeletal and connective tissue disorders) | 8 | 5 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 5 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 19 | 9 | 10
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 11 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 16 | 12 | 12
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 21 | 14 | 10
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
Dizziness (Nervous system disorders) | 10 | 9 | 8
Headache (Nervous system disorders) | 29 | 28 | 20
Hypoaesthesia (Nervous system disorders) | 8 | 6 | 7
Migraine (Nervous system disorders) | 1 | 6 | 5
Paraesthesia (Nervous system disorders) | 7 | 8 | 3
Depression (Psychiatric disorders) | 5 | 7 | 4
Insomnia (Psychiatric disorders) | 5 | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 19 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 21 | 12 | 7
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 4
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 | 6 | 4
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 6 | 5
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Eczema (Skin and subcutaneous tissue disorders) | 5 | 5 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Night Sweats (Skin and subcutaneous tissue disorders) | 4 | 8 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 7 | 7
Rash (Skin and subcutaneous tissue disorders) | 17 | 16 | 8
Hypertension (Vascular disorders) | 14 | 15 | 6

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <= 5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.